CLINICAL TRIAL: NCT02524210
Title: Effect of Inhibitors of the Proton Pump on Intestinal Transporters and Their Impact on the Pharmacokinetics of Dabigatran - Mechanistic and Clinical Approach -BIPP Study
Brief Title: Effect of Inhibitors of the Proton Pump on Intestinal Transporters
Acronym: BIPP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: 1208088; 2013-004932-31 (EudraCT Number); 140096A-21 (Other: ANSM)
Record Dates: First submitted 2015-08-13; First posted 2015-08-14 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: volunteers
MeSH Terms: interventions — Dabigatran; Rabeprazole; Omeprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Experimental): * Period " Dabigatran"
  * Washout period (at least 6 days)
  * Period " Rabeprazole + Dabigatran"
  * Washout period (at least 6 days)
  * Period " Omeprazole + Dabigatran"
  Interventions: Drug: Dabigatran; Drug: Rabeprazole and Dabigatran; Drug: Omeprazole and Dabigatran
- Arm B (Experimental): * Period "Rabeprazole + Dabigatran "
  * Washout period (at least 6 days)
  * Period " Dabigatran"
  * Washout period (at least 6 days)
  * Period " Omeprazole + Dabigatran"
  Interventions: Drug: Dabigatran; Drug: Rabeprazole and Dabigatran; Drug: Omeprazole and Dabigatran
- Arm C (Experimental): * Period " Rabeprazole + Dabigatran"
  * Period " Omeprazole + Dabigatran"
  * Period " Dabigatran"
  Interventions: Drug: Dabigatran; Drug: Rabeprazole and Dabigatran; Drug: Omeprazole and Dabigatran

INTERVENTIONS:
Drug: Dabigatran — dabigatran etexilate 150 mg/day (1 day)
Drug: Rabeprazole and Dabigatran — rabeprazole 20 mg / day for 5 days, then the 6th day concomitant rabeprazole 20 mg of dabigatran etexilate 150 mg;
Drug: Omeprazole and Dabigatran — omeprazole 20 mg / day for 5 days, then the sixth day concomitant omeprazole 20 mg and 150 mg dabigatran etexilate

SUMMARY:
Dabigatran etexilate is a novel oral anticoagulant. It is indicated in venous thromboembolic prevention in orthopedic surgery and has recently shown greater efficiency and tolerance as anticoagulants in preventing thromboembolism in atrial fibrillation. However, it increases the risk of gastrointestinal bleeding compared to standard treatment (AVK) [3]. In these circumstances the risk / benefit of dabigatran could be improved by combining it with gastric protectors such as inhibitor drugs proton pump (IPP).

Investigators want to evaluate the pharmacokinetic and pharmacodynamic effects of co-administration of these two IPP (omeprazole, rabeprazole) with dabigatran in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* weight between 60 and 85 kg
* normal clinical exam
* normal biological exam

Exclusion Criteria:

* hypersensitivity to dabigatran or any of its excipients
* hypersensitivity to omeprazole or rabeprazole or any of its excipients
* previous history of hemorrhagic disease
* insufficiency liver
* severe kidney failure
* peptic ulcer
* Any drug taken during the week before the start of the study
* smoker
* Consumption of grapefruit juice
* practice of violent sport

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) from plasma concentrations of dabigatran | baseline after each dose of dabigatran etexilate.
  Area under the curve (AUC) from plasma concentrations of dabigatran
Area under the curve (AUC) from plasma concentrations of dabigatran | 0.25 hours after each dose of dabigatran etexilate.
Area under the curve (AUC) from plasma concentrations of dabigatran | 0.5 hours after each dose of dabigatran etexilate.
Area under the curve (AUC) from plasma concentrations of dabigatran | 1 hour after each dose of dabigatran etexilate.
Area under the curve (AUC) from plasma concentrations of dabigatran | 1.5 hours after each dose of dabigatran etexilate.
Area under the curve (AUC) from plasma concentrations of dabigatran | 2 hours after each dose of dabigatran etexilate.
Area under the curve (AUC) from plasma concentrations of dabigatran | 3 hours after each dose of dabigatran etexilate.
Area under the curve (AUC) from plasma concentrations of dabigatran | 6 hours after each dose of dabigatran etexilate.
Area under the curve (AUC) from plasma concentrations of dabigatran | 8 hours after each dose of dabigatran etexilate.
Area under the curve (AUC) from plasma concentrations of dabigatran | 12 hours after each dose of dabigatran etexilate.
Area under the curve (AUC) from plasma concentrations of dabigatran | 24 hours after each dose of dabigatran etexilate.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BERTOLETTI, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France